CLINICAL TRIAL: NCT02944708
Title: A Randomized Phase III Trial Evaluating Maintenance Chemotherapy for Metastatic Nasopharyngeal Carcinoma
Brief Title: Trial Evaluating Maintenance Chemotherapy for Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Collaborators: Fudan University (Other); Eye & ENT Hospital of Fudan University (Other); The First Affiliated Hospital of Xiamen University (Other); Jiangxi Provincial Cancer Hospital (Other); Taichung Veterans General Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Cancer Hospital of Guangxi Medical University (Other); National Cancer Centre, Singapore (Other); West China Hospital (Other); Peking University Cancer Hospital & Institute (Other); Tongji Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Lin Kong, Consultant doctor, chair of head and neck cancer, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2015-04
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: maintenance chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conventional chemotherapy (Active Comparator): Patients in this arm will only receive 4-8 cycles of cisplatin-based regimen. TPF ( docetaxel, cisplatin and 5-fluorouracil ), TP (docetaxel and cisplatin), GP (gemcitabine and cisplatin) and PF (cisplatin and 5-fluorouracil) regimens are preferred.
  Interventions: Drug: Conventional chemotherapy
- Maintenance chemotherapy 1 (Experimental): Patients in this arm will receive 6 cycles of oral fluoropyrimidine monotherapy as maintenance therapy, in addition to 4-8 cycles of cisplatin-based standard chemotherapy.
  Interventions: Drug: Conventional chemotherapy; Drug: Maintenance chemotherapy 1
- Maintenance chemotherapy 2 (Experimental): Patients in this arm will receive oral fluoropyrimidine maintenance therapy until disease progression or intolerable toxicities, after 4-8 cycles of cisplatin-based standard chemotherapy.
  Interventions: Drug: Conventional chemotherapy; Drug: Maintenance chemotherapy 2

INTERVENTIONS:
Drug: Conventional chemotherapy
Drug: Maintenance chemotherapy 1
  Arms: Maintenance chemotherapy 1
Drug: Maintenance chemotherapy 2
  Arms: Maintenance chemotherapy 2

SUMMARY:
The purpose of this study is to examine the efficacy of maintenance chemotherapy for the treatment of metastatic nasopharyngeal carcinoma. Participants will be randomized to 3 arms. Arm 1, control group, participants will receive only 4-8 cycles of conventional chemotherapy; arm 2, participants will receive 6 cycles of maintenance chemotherapy after conventional chemotherapy; arm 3, experiment arm, after conventional chemotherapy, participants will receive maintenance chemotherapy until disease progression or intolerable toxicities.

DETAILED DESCRIPTION:
This is a phase 3 randomized clinical trial to determine the efficacy of maintenance chemotherapy for the treatment of metastatic chemotherapy and how it should be delivered. Participants will be randomized to 3 arms. Arm 1 (control group), participants will receive only conventional chemotherapy; arm 2 (experimental group), participants will receive up to 6 cycles of maintenance chemotherapy after conventional chemotherapy; arm 3 (experimental group), after conventional chemotherapy, participants will receive maintenance chemotherapy until disease progression or intolerable toxicities. Participants in all 3 arms will receive similar conventional chemotherapy. Four to eight cycles of conventional chemotherapy with platinum-based regimen is preferred. Maintenance chemotherapy should use one of the regimens: S1 (40mg, twice a day for 14 days, every 3 weeks), capecitabine (1000mg/m^2, twice a day for 14 days, every 3 weeks) or Tegafur-uracil (100mg/m^2, q8h, for 14 days, every 3 weeks). The response of treatment will be evaluated according to RECIST criteria. Adverse events will be documented according to CTCAE v4.03.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 70 years
* Histologically confirmed nasopharyngeal carcinoma, WHO (World Health Organization) classification II/III
* With distant metastasis
* With measurable lesions that can be detected by imaging studies
* Achieving PR (partial response) after 4 cycles of conventional chemotherapy
* Life expectancy ≥ 6 months
* ECOG (Eastern Cooperative Oncology Group): 0-1, no significant active concurrent medical illnesses
* Adequate laboratory values within 30 dyas of enrollment to study defined as follows: N > 2000/mm^3; PLT (platelet count) > 100,000/mm^3; total bilirubin < 1.5mg/dl; AST (aspartate aminotransferase)/ALT (alanine aminotransferase) < 1.5 ULN (upper limit of normal); SCr (serum creatinine) < 1.5mg/dl; CCR (creatinine clearance rate) > 60ml/min
* Willing to accept adequate contraception for women with childbearing potential
* Ability to understand character and individual consequences of the clinical trial
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial

Exclusion Criteria:

* Received previous treatment for metastatic disease
* Pregnant or lactating women
* A diagnosis of malignancy other than CIS (carcinoma in situ) of the cervix, BCC (basal cell carcinoma) and SCC (squamous cell carcinoma) of the skin within the past 5 years
* Refusal of the patient to participate into the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From the time point the patients are included in the study, median of 3 years.

SECONDARY OUTCOMES:
Overall survival | From the time point the patients are included in the study, median of 3 years.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | From the time point the patients are included in the study, median of 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jiade J Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center,Shanghai, SPHIC
Locations (14):
- China (12):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Jiangxi Province Tumor Hospital, Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer center, Shanghai, Shanghai Municipality
  - Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality
  - Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Chengdu, Sichuan
- National Cancer Centre, Singapore, Singapore, Singapore
- Taichung Veterans General Hospital, Taichung, Taiwan